CLINICAL TRIAL: NCT01804179
Title: Colorectal Cancer Awareness, Research, Education and Screening (CARES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-16447
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: colon; rectum; cancer; screening; questionnaire; testing; educational materials
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Intervention (SI) (Active Comparator): At Baseline Visit, Participants in the standard intervention (SI) condition will get: I-FOBT kit and "Screen for Life" brochure, a mailed reminder card at two weeks post-intervention to remind them about FOBT testing and follow up assessments at 12 months.
  Interventions: Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit; Other: Standard Intervention (SI) Educational Materials; Other: Baseline Visit Survey; Other: Follow-up Questionnaire
- CARES Intervention (Experimental): Colorectal Cancer Awareness, Research, Education and Screening (CARES). At Baseline Visit, Participants in the CARES intervention will receive: I-FOBT kit, a newly developed DVD and booklet, and a mailed reminder card at two weeks post-intervention to remind them about FOBT testing, and follow-up assessments at 12 months.
  Interventions: Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit; Other: CARES Intervention Educational Materials; Other: Baseline Visit Survey; Other: Follow-up Questionnaire

INTERVENTIONS:
Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit — Participants will receive an Immunochemical Fecal Occult Blood Test (I-FOBT) Kit (a home stool blood test) used as a first-step screening tool for colorectal cancer to take home. The research staff will provide instructions on how to use the kit.
  Other Names: Home Stool Blood Test; fecal immunochemical test (FIT)
Other: Standard Intervention (SI) Educational Materials — "Screen for Life" brochure
  Arms: Standard Intervention (SI)
Other: CARES Intervention Educational Materials — Newly developed digital video disc (DVD) and booklet
  Arms: CARES Intervention
Other: Baseline Visit Survey — In both conditions, patients will participate in a Baseline Survey. Three brief items will be used to assess patient-provider discussion and recommendation: (1) Was colorectal cancer or colorectal cancer screening one of the things you discussed with the doctor or health care provider? (Yes/No). (2) If Yes, who brought the topic of colorectal cancer first? (patient/health care provider). (3) Did your doctor or health care provider recommend colorectal cancer screening? (Yes/No). These questions are necessary to evaluate the impact of interventions on patient-provider discussion of CRCS and provider recommendation of CRCS.
Other: Follow-up Questionnaire — 12 months after participants began to participate in the study, they will be contacted via telephone to complete a final set of questionnaires. Participants will be asked questions similar to those answered in baseline. This time they will ask about the participant's thoughts on the educational materials as well.

SUMMARY:
There are two parts to this study: (1) an information gathering phase leading to the development of new educational materials; and (2) a study to test the newly developed material. The information gathering phase has been completed. The purpose of this part of the research study is to test the usefulness and acceptability of new educational materials investigators have developed. Investigators will compare the new educational material to another widely available educational brochure. The goal is to see if the new educational material will change knowledge and behaviors about colorectal cancer and colorectal screening.

DETAILED DESCRIPTION:
Federally qualified health centers (FQHCs) and other community health clinics (CHCs) provide comprehensive primary health care for underserved patients. Recently, high-sensitivity and high-specificity fecal occult blood tests (FOBT) and fecal immunochemical tests (FIT) have emerged as a preferred initial screening modality within clinics due to convenience, ease of use, and low cost compared with colonoscopy. FOBT/FIT may help to reduce colorectal cancer screening (CRC) screening disparities and overcome several previously mentioned factors that often account for suboptimal CRC screening rates.

ELIGIBILITY:
Inclusion Criteria:

* Racially-ethnically diverse adult men and women
* Average risk individuals who have no personal diagnosis, or presumptive symptoms of colorectal cancer (CRC), or are not at high risk
* Self-report as not current on screening
* Provide at least two forms of contact information and contact information of a relative (not living with respondent) to facilitate follow-up contacts
* Are able to speak, read and write English because the instruments and CARES intervention are available only in English at this time. We recognize that interventions are needed for non-English speaking populations, therefore, once we find promise in the English language CARES intervention materials, we will move forward with conducting other studies that involve translation of measures and cultural adaptation of the CARES intervention materials into Spanish or Haitian Creole.

Exclusion Criteria:

* Individuals who have participated in a CRCS research study in the past 1 year will not be eligible for this study.
* Recent screening criteria relates to not having had I-FOBT within the previous year, flex sig within the previous 5 years, a double-contrast barium enema (DCBE) x-ray with the previous 5 years, or a colonoscopy within the previous 10 years.
* Within the recruitment and intervention frame, high risk individuals (due to strong family history, ulcerative colitis, polyposis syndromes) are excluded because they may be eligible for CRC screening before age 50, and the preferred screening option is certainly colonoscopy which is beyond the primary focus of the current study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Rate of Test Kit Completion | 6 months post final enrollment
  Investigators will measure uptake of I-FOBT/FIT as any completed kit within 180 days of delivery of the intervention. That is, the proportion of participants who return a sampled kit by the 6 month assessment (investigators expect most kits to be returned much sooner) for calculation of the primary screening endpoint. I-FOBT/FIT use will be compared (CARES vs. SI).

SECONDARY OUTCOMES:
Overall Colorectal Cancer Screening (CRCS) With Any Test | 12 months post final enrollment
  Overall CRCS with any test will be compared (CARES vs. SI). It is expected that pairing I-FOBT/FIT kits with the CARES toolkit will result in greater CRCS uptake compared to SI plus I-FOBT/FIT.
Time to Kit Return | Up to 12 months post final enrollment
  Maximum number of months required for kit return per study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Gwede, PhD, MPH, RN, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: A Randomized Controlled Trial of a Multicomponent, Targeted, Low-Literacy Educational Intervention Compared With a Nontargeted Intervention to Boost Colorectal Cancer Screening With Fecal Immunochemical Testing in Community Clinics — http://onlinelibrary.wiley.com/doi/10.1002/cncr.30481/full